CLINICAL TRIAL: NCT00629655
Title: A Spinal fMRI Study of Resting-State, Motor Task and Acupoint Stimulation
Brief Title: A Spinal Functional Magnetic Resonance Imagine (fMRI) Study of Resting-State, Motor Task and Acupoint Stimulation
Status: Completed | Type: Observational
Sponsor: China Rehabilitation Research Center (Other Government)
Collaborators: Ministry of Finance, China (Other Government); Capital Medical University (Other)
Responsible Party: Pengxu Wei, China Rehabilitation Research Center
Other Study IDs: 2007CZ-4
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Cerebral Infarction
Keywords: fMRI; spinal cord; human; health; cerebral infarction; healthy
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: healthy people, male
  Interventions: Other: motor task, sensory stimulation
- 2: male patients with cerebral infarction, chronic stage
  Interventions: Other: motor task, sensory stimulation

INTERVENTIONS:
Other: motor task, sensory stimulation — motor task: finger tapping, simple type and complex type
  sensory stimulation: electric or tactile stimulation
  Other Names: group 1:healthy people; group 2:patients with cerebral infarction,chronic stage

SUMMARY:
The spinal cord is a very important part of the central nervous system. fMRI can be applied to observe functional status of the human spinal cord. Under different conditions, the investigators will see different types of fMRI signals within the spinal cord. In resting state, the investigators might see active/inactive signals, too.

ELIGIBILITY:
Inclusion Criteria (for healthy people):

* Chinese male residents
* right handed
* no history of psychological/psychotic problems
* no history of important diseases

Exclusion Criteria (for healthy people):

* with factors which make subjects unsuitable to receive MR examination
* history of important diseases

Inclusion Criteria (for patients):

* Chinese male patients with ischemic stroke (CT/MRI scan confirmed)
* right handed
* at least 1.5 months from onset of stroke
* ability to follow complex commands

Exclusion Criteria (for patients):

* hemodynamic instability
* history of dementia
* inability to give consent because of impaired cognition or receptive aphasia
* diseases in spine/spinal cord
* with factors which make subjects unsuitable to receive MR examination

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: group 1: male residents of Beijing group 2: male stroke patients of Beijing Boai hospital
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
fMRI | one day

CONTACTS AND LOCATIONS:
Overall Officials: Pengxu Wei, Master, Principal Investigator — China Rehabilitation Research Center
Locations (1):
- Beijing Boai Hospital, Beijing, Beijing Municipality, China